CLINICAL TRIAL: NCT05160675
Title: Nutrition, Microbiome and Bone Health During Early Life Related to Health
Acronym: Bamboo
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Tianjin Women and Children's Health Center (Other); BGI-research (Other); Cognizant Technology Solutions AG (Unknown); SAS Institute (Industry); Veeva Systems (Industry)
Responsible Party: Sponsor
Other Study IDs: 20.27.NRC
Record Dates: First submitted 2021-10-13; First posted 2021-12-16 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fecal, urine sample of the infants, and breastmilk from the mothers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Group 1: 690 healthy infants and their mother followed from birth to 12 months
- Group 2: Group 2: 690 healthy infants and their mother followed from 6 months to 3 years of age

INTERVENTIONS:
Other:  — No intervention

SUMMARY:
The aim of the study is to establish the longitudinal microbiome and bone trajectories from birth to 3 years, and to evaluate the influence of nutrition on these trajectories.

DETAILED DESCRIPTION:
The main objective of the study is to understand the influence of nutrition and dietary patterns on microbiome and bone trajectories during early life. Specific research objectives are:

* Establish the reference trajectories of gut microbiome maturation index and bone development in healthy Chinese children aged 0-3years
* Assess the impact of early life nutrition on gut microbiome trajectory
* Investigate the influence of microbiome, early life parameters and nutritional parameters on bone health

ELIGIBILITY:
Inclusion Criteria:

* It is important to carefully consider whether a subject is suitable for enrollment into this observational study. Fulfillment of the inclusion and exclusion criteria for each subject will be documented by a qualified member of the investigative staff before any subject is enrolled.

Healthy infants who fulfill all the following inclusion criteria will be included:

1. Having obtained his/her parents' (or his/her legally accepted representative's [LAR's]) written informed consent and having evidence of personally signed and dated informed consent document indicating that the subject's parents/LAR have been informed of all pertinent aspects of the study.
2. Subject's parent(s)/LAR is of legal age of consent, is willing and able to fulfill the requirements of the study protocol.
3. For group 1, healthy infants aged ≤ 10 days after birth (date of birth = Day 0).

   For group 2, healthy infants with maximum age of 6 months
4. Full-term gestational birth (≥ 37 and ≤ 42 weeks).
5. Subject's parent(s)/LAR is able to be contacted directly by telephone throughout the study.
6. Both parents registered have a fixed work and / or residence within their jurisdiction.

Exclusion Criteria:

1. Complicated pregnancy (e.g., preeclampsia, gestational diabetes, bowel disease) as assessed by medical interview/ medical record when available
2. Infant's parents/LAR not willing and/or not able to comply with scheduled visits and the requirements of the study protocol
3. Currently participating or having participated in another clinical trial within 4 weeks prior to trial start.

Ages: 0 Days to 6 Months | Sex: All
Age Groups: Child
Study Population: Group 1: 690 healthy infants and their mother followed from birth to 12 months Group 2: 690 healthy infants and their mother followed from 6 months to 3 years of age
Sampling Method: Non-Probability Sample
Enrollment: 2760 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
gut microbiome | Group 1: 0-1 year, Group 2: 0.5-3 years
  microbiome maturation index derived from microbial composition, bacteria function, metabolites
dietary factors | Group 1: 0-1 year, Group 2: 0.5-3 years
  derived from infant questionnaires
dietary factors | Group 1: 0-1 year, Group 2: 0.5-3 years
  derived from food diaries of the types of complementary feeding, the food consumption, the nutrient intakes, the food source of nutrients, the dietary patterns
bone development | Group 1: 0-1 year, Group 2: 0.5-3 years
  bone tibia speed of sounds (SOS) (meter / second) using ultrasound
bone health | Group 1: 0-1 year, Group 2: 0.5-3 years
  Bone tibia length using ruler (cm)
dietary intakes and health outcomes | Group 1: 0-1 year, Group 2: 0.5-3 years
  derived from infant questionnaires and their food diaries of the types of complementary feeding, the food consumption, the nutrient intakes, the food source of nutrients, the dietary patterns

SECONDARY OUTCOMES:
Gut microbiome | Group 1: 0-1 year, Group 2: 0.5-3 years
  microbiome maturation index derived from microbial composition, bacteria function, metabolites
Urinary markers of bone metabolism | Group 1: 0-1 year, Group 2: 0.5-3 years
  urinary resorption biomarkers which are Pyridinolin and Deoxypiridinolin Crosslinks by ELISA
breast milk composition | Group 1: 0-3 months
  breast milk composition, macro and micronutrients (e.g. protein, mineral, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Gongshu Liu, Dr., Principal Investigator — Tianjin Women and Children Health Center
Locations (1):
- Tianjin Women and Children Health Center，, Tianjin, China

IPD SHARING:
Plan to Share IPD: No